CLINICAL TRIAL: NCT02414295
Title: Management of Azoospermic Patients With Kleinfelter Syndrome Patients With Mesenchymal Stem Cell Injection
Brief Title: Sperm Production in Kleinfelter Syndrome Patients After Mesenchymal Stem Cell Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Man Clinic for Andrology, Male Infertility and Sexual Dysfunction (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 6714
Record Dates: First submitted 2014-08-21; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Klinefelter Syndrome; Azoospermia
Keywords: Stem cell; Kleinfelter syndrome; Azoospermia; Sterility; Infertility
MeSH Terms: conditions — Klinefelter Syndrome; Azoospermia; Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stem cell injection (Experimental): Bone marrow Mesenchymal stem cell injection in the testicular tubules and testicular artery
  Interventions: Drug: Mesenchymal stem cell injection

INTERVENTIONS:
Drug: Mesenchymal stem cell injection — Aspirated bone marrow then separation for Mesenchymal stem cell

SUMMARY:
Klinefelter syndrome KS is caused by an additional X chromosome in males (47,XXY). Clinical findings are nonspecific during childhood; thus, the diagnosis commonly is made during adolescence or adulthood in males who have small testes with hypergonadotropic hypogonadism and gynecomastia. Virtually all men with Klinefelter syndrome are infertile.

Approximately one in 1,000 boys is born with an additional X chromosome-47,XXY, the karyotype that causes Klinefelter syndrome. This karyotype is detected at or before birth in 10 percent of affected boys, and it is found during adulthood in 25 percent of affected men. Almost all men with a 47,XXY karyotype will be infertile; Klinefelter syndrome accounts for 3 percent of male infertility.

Klinefelter syndrome is common in infertile men with oligospermia or azoospermia (5 to 10 percent).

Infertility in men with Klinefelter syndrome is caused by a precipitous drop in sperm count. If sperm are present, cryopreservation is useful for future family planning with intracytoplasmic sperm injection, and if not, testicular sperm extraction may be pursued. Although there have been multiple reports of successful fertilization by men with Klinefelter syndrome.

Mesenchymal stem cell injection in testicular tubules and intra testicular artery using surgical microscope.

The period for follow up last from three months to twelve months including semen analysis to detect sperm and hormonal profile .

DETAILED DESCRIPTION:
The problem started with this kind of patinets when underwent multiple TESE without sperm.

The investigators try to inject KS patients with mesenchymal stem cells to stimulate testicular tissue for production of sperms.

before injection the investigators measure:( FSH, LH, Testosterone, Prolactin, Inhibin B, Karyotyping, Azoospermic Factor, Testicular size by ultrasound).

Three to twelf months after stem cell injection the investigators reevaluate patients by the same measure to demoenstarte any changes.

ELIGIBILITY:
Inclusion Criteria:

* Kleinfelter syndrome
* Azoospermia
* Negative TESE

Exclusion Criteria:

* Absent Testes

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sperm detection | 12 months
  Semen Analysis

SECONDARY OUTCOMES:
Hormonal profile | 12 months
  Inhibine B, FSH, LH

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Gadalla, MD, Principal Investigator — Al-Azhar University
Locations (1):
- Man Clinic for Andrology and male infertility, Cairo, Egypt